CLINICAL TRIAL: NCT03970031
Title: MMONARCh-1: Study of MSDC-0602K, a Modulator of the Mitochondrial Pyruvate Carrier for Outcomes in Patients With Pre Type 2 Diabetes (T2D) or T2D and NAFLD/NASH, Assessed for ImpRoved Glycemic Control and Cardiovascular Outcomes-1
Brief Title: A Study of MSDC-0602K to Assess Glycemic Control and Cardiovascular Outcomes in Patients With Pre-T2D or T2D and NAFLD/NASH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cirius Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTI-0602K-C013
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Type2 Diabetes; NASH - Nonalcoholic Steatohepatitis; Nonalcoholic Steatohepatitis; Non-Alcoholic Fatty Liver Disease
Keywords: Diabetes; NASH; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MSDC-0602K (Active Comparator): MSDC-0602K one tablet per day taken orally
  Interventions: Drug: MSDC-0602K
- Placebo (Placebo Comparator): Placebo one tablet per day taken orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MSDC-0602K — MSDC-0602K tablet
  Arms: MSDC-0602K
Drug: Placebo — Matching tablet
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind study of MSDC-0602K or placebo in subjects with pre-T2D or T2D and evidence of NAFLD/NASH.

DETAILED DESCRIPTION:
This is a randomized, double-blind study of MSDC-0602K or placebo given orally once daily to subjects with pre-T2D or T2D and evidence of NAFLD/NASH. Visits will include a Screening Period, a minimum Treatment of 26 weeks, and a Long-Term Follow-up Period during which subjects will continue taking assigned treatment.

Safety will be assessed by periodic measurement of vital signs, physical examinations, blood laboratory analyses, and the occurrence of adverse events.

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent.
2. Adult subjects with an age of > 18 years but < 80 years.
3. Male or female subjects with reproductive potential must agree to comply with approved double barrier contraceptive method for the duration of the trial. Females of non-childbearing potential are considered:

   Post-menopausal Surgically sterile
4. Diagnosis of NAFLD
5. AST>27 U/L
6. HgbA1c >6%
7. Diagnosis of Pre-T2D or T2D
8. History of macrovascular cardiovascular disease

Key Exclusion Criteria:

1. Prior liver transplantation or currently on transplant list.
2. Other well-documented causes of active chronic liver disease
3. Current cirrhosis
4. Pregnant or nursing women
5. AST or ALT > 5 times the upper limit of normal
6. Total bilirubin > 1.3 mg/dL unless diagnosis of Gilbert's disease with direct bilirubin within normal reference range
7. Serum albumin < 3.5 g/dL at Screening
8. Alkaline phosphatase >2 times the upper limit of normal at Screening
9. Estimated glomerular filtration rate (eGFR by MDRD) <30 ml/min/1.73 m2 but ≤75 ml/min/1.73 m2
10. In patients who are not anticoagulated, INR ≥ 1.3 times ULN at Screening or other evidence of impaired coagulation.
11. Acute vascular events including ACS, stroke or TIA, worsening of peripheral vascular disease or any vascular/cardiac procedure
12. Limb amputation for reason other than trauma.
13. HbA1c >10%
14. Any planned surgery or device implantation after screening
15. Ejection fraction < 35% or Heart failure with NYHA class IV
16. History of alcohol abuse or drug abuse within 6 months prior to Screening Diagnosis at any time of Type 1 diabetes.
17. Current or history of recent (≤ 6 months) use of ursodeoxycholic acid.
18. Current use of insulin.
19. Current use of thiazolidinediones.
20. Any history or current concomitant disorder such as haematological, pulmonary, metabolic, endocrine disorders that are severe or life-threatening.
21. Use of concomitant medications with a known significant metabolism by CYP2C8 including paclitaxel or repaglinide for the duration of the study.
22. History of diabetic ketoacidosis or hyperosmolar non-ketotic coma within the 6 months prior to Screening.
23. Known or suspected intolerance or hypersensitivity to the study drugs, closely related compounds such as PPARγ agonists (pioglitazone or rosiglitazone), or any of their stated ingredients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in glycosylated hemoglobin (HbA1c) from baseline to Week 26 | 26 weeks
Change in the weighted average of standardized AST, CK-18, and HbA1c values (standard deviations) from baseline to Week 26 | 26 weeks
  This is a single composite outcome measure. This is derived by standardizing the values of AST, CK-18, and HbA1c by subtracting the respective study population means and dividing by respective study population standard deviations at each time point; averaging these standardized AST, CK-18,and HbA1c values (or z-scores) for a given patient at each time point; and then computing the difference from baseline to week 26 with respect to these averages.

SECONDARY OUTCOMES:
Time to first event of death, adjudicated nonfatal MI or USA hospitalization, adjudicated hospital admission for HF, or adjudicated nonfatal ischemic stroke. | through study completion, an expected average of 15 months
Time to first event of death or adjudicated non-fatal MI or USA hospitalization, adjudicated hospital admission for HF, adjudicated nonfatal ischemic stroke, or liver event in all randomized subjects. | through study completion, an expected average of 15 months
  A liver event consists of ascites (confirmed by paracentesis or abdominal imaging), hepatic encephalopathy (defined clinically), variceal hemorrhage (confirmed by endoscopy), or liver transplant.

IPD SHARING:
Plan to Share IPD: No